CLINICAL TRIAL: NCT01386385
Title: A Dose Finding Study Followed by Phase II Randomized, Placebo-Controlled Study of Veliparib (ABT-888) Added to Chemoradiotherapy With Carboplatin and Paclitaxel for Unresectable Stage III Non-small Cell Lung Cancer (NSCLC), (NCI Study Number 8811)
Brief Title: Veliparib With or Without Radiation Therapy, Carboplatin, and Paclitaxel in Patients With Stage III Non-small Cell Lung Cancer That Cannot Be Removed by Surgery
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NCI-2011-02592; NCI-2011-02592 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CHNMC-PHII-111; CDR0000701003; PHII-111; S1206; 8811 (Other: SWOG); 8811 (Other: CTEP); N01CM62209 (NIH); U10CA032102 (NIH); U10CA180888 (NIH)
Record Dates: First submitted 2011-06-30; First posted 2011-07-01 (Estimated); Results first posted 2021-07-12 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-10

CONDITIONS: Lung Adenocarcinoma; Lung Adenocarcinoma, Mixed Subtype; Lung Large Cell Carcinoma; Lung Squamous Cell Carcinoma; Minimally Invasive Lung Adenocarcinoma; Stage III Lung Non-Small Cell Cancer AJCC v7; Stage IIIA Lung Non-Small Cell Cancer AJCC v7; Stage IIIB Lung Non-Small Cell Cancer AJCC v7
MeSH Terms: conditions — Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar | interventions — Radiotherapy, Conformal; Carboplatin; Paclitaxel; Taxes; veliparib

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (RT, veliparib, carboplatin, paclitaxel) (Experimental): Patients undergo 3D-CRT and receive veliparib, carboplatin, and paclitaxel as in Phase I induction and consolidation therapy.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Drug: Carboplatin; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Drug: Veliparib
- Arm II (3D-CRT, placebo, carboplatin, paclitaxel) (Active Comparator): Patients undergo 3D-CRT as in arm I. Patients also receive placebo PO BID on days 1-43 and carboplatin and paclitaxel as in Phase I. Within 4-6 weeks after completion of chemotherapy and radiation therapy, patients receive placebo on days 1-7 and carboplatin and paclitaxel as in Phase I.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Drug: Carboplatin; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Other: Placebo Administration

INTERVENTIONS:
Radiation: 3-Dimensional Conformal Radiation Therapy — Undergo 3D-conformal RT
  Other Names: 3-dimensional radiation therapy; 3D Conformal; 3D CONFORMAL RADIATION THERAPY; 3D CRT; 3D radiotherapy; 3D-CRT; Conformal Therapy; Radiation Conformal Therapy; Radiation, 3D Conformal; Three dimensional external beam radiation therapy (procedure)
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Other: Placebo Administration — Given PO
  Arms: Arm II (3D-CRT, placebo, carboplatin, paclitaxel)
Drug: Veliparib — Given PO
  Other Names: ABT 888; ABT-888; ABT888; PARP-1 inhibitor ABT-888
  Arms: Arm I (RT, veliparib, carboplatin, paclitaxel)

SUMMARY:
This phase I/II partially randomized trial studies the side effects and best dose of veliparib when given together with radiation therapy, carboplatin, and paclitaxel and to see how well it works in treating patients with stage III non-small cell lung cancer that cannot be removed by surgery. Veliparib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Drugs used in chemotherapy, such as carboplatin and paclitaxel, work in different ways to stop the growth of tumor cells either by killing the cells, by stopping them from dividing, or by stopping them from spreading. It is not yet known whether radiation therapy, carboplatin, and paclitaxel are more effective with or without veliparib in treating non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish the maximum tolerated dose (MTD) and the recommended phase II dose of ABT-888 (veliparib) when given concurrently with standard carboplatin/paclitaxel and radiotherapy in patients with unresectable stage III non-small cell lung cancer (NSCLC). (Phase I) II. To assess whether carboplatin/paclitaxel plus ABT-888 compared with carboplatin/paclitaxel plus placebo improves progression-free survival (PFS) in patients with unresectable stage III NSCLC. (Phase II) III. To compare overall survival (OS) in patients treated with carboplatin/paclitaxel and radiotherapy plus ABT-888 to those treated with carboplatin, paclitaxel and radiotherapy plus placebo. (Phase II) IV. To assess the response rate (confirmed and unconfirmed, complete and partial responses) and disease control rate in the subset of patients with measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) criteria. (Phase II) V. To assess the safety and toxicity profile of the regimen. (Phase II)

SECONDARY OBJECTIVES:

I. To collect tumor tissue from pretreatment biopsies (archival samples) for biomarker studies, including poly (ADP-ribose) polymerase 1 (PARP) activity by measuring the levels of poly-ADP-ribose, gamma-H2A histone family, member X (gamma-H2AX), and messenger ribonucleic acid (mRNA) expression levels of deoxyribonucleic acid (DNA) repair enzymes such as excision repair cross-complementing rodent repair deficiency, complementation group 1 (ERCC1)/x-ray repair complementing defective repair in Chinese hamster cells 1 (XRCC1).

II. To collect blood samples for evaluation of gamma-H2AX (circulating tumor cells) and other relevant future studies.

OUTLINE: This is a phase I, dose-escalation study of veliparib followed by a randomized phase II study.

PHASE I:

INDUCTION THERAPY: Patients undergo 3-dimensional conformal radiation therapy (3D-CRT) once daily (QD), 5 days a week, for 6 weeks. Patients also receive veliparib orally (PO) twice daily (BID) on days 1-43 and carboplatin intravenously (IV) over 30 minutes and paclitaxel IV over 1 hour on days 1, 8, 15, 22, 36, and 43 in the absence of disease progression or unacceptable toxicity. Patients without disease progression after completion of chemoradiotherapy undergo consolidation therapy.

CONSOLIDATION THERAPY: Beginning within 4-6 weeks of chemotherapy and radiation therapy, patients receive veliparib PO BID on days 1-7 (course 1) and 22-28 (course 2) and carboplatin IV over 30 minutes and paclitaxel IV over 3 hours on day 1 and on day 22 of course 2. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity.

PHASE II: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients undergo 3D-CRT and receive veliparib, carboplatin, and paclitaxel as in Phase I induction and consolidation therapy.

ARM II: Patients undergo 3D-CRT as in arm I. Patients also receive placebo PO BID on days 1-43 and carboplatin and paclitaxel as in Phase I. Within 4-6 weeks after completion of chemotherapy and radiation therapy, patients receive placebo on days 1-7 and carboplatin and paclitaxel as in Phase I.

After completion of study treatment, patients are followed up every 4 months for first 2 years and then every 6 months until 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically-proven new diagnosis of unresectable stage IIIA/IIIB*, non-small cell lung cancer (adenocarcinoma, bronchioloalveolar cell carcinoma, large cell carcinoma, squamous cell carcinoma, or mixed)

  * Per the American Joint Committee on Cancer (AJCC) 7th edition, pleural and pericardial are now considered stage M1a disease; when pleural fluid is visible on the computed tomography (CT) scan or on a chest x-ray, a thoracentesis is required to confirm that the pleural fluid is cytologically negative; patients with exudative pleural effusions are excluded, regardless of cytology; patients with effusions that are minimal (i.e. not visible on chest x-ray) that are too small to safely tap are eligible; a small effusion that has positive fludeoxyglucose F 18 (FDG) uptake on positron emission tomography (PET) has to be proven to be malignant per standard of care diagnostic procedures for the patient to be excluded
* Patients must have measurable or non-measurable disease documented by CT, magnetic resonance imaging (MRI) or PET/CT; the CT from a combined PET/CT may be used to document only non-measurable disease unless the scan is of diagnostic quality; measurable disease must be assessed by CT within 28 days prior to registration; pleural effusions, ascites and laboratory parameters are not acceptable as the only evidence of disease; non-measurable disease must be assessed within 42 days prior to registration; all disease must be assessed and documented on the Baseline Tumor Assessment Form
* Patients with brain metastases are ineligible; all patients must have a pretreatment CT or MRI scan of the brain to evaluate for central nervous system (CNS) disease within 42 days prior to registration
* Patients must not have received any prior systemic therapy (chemotherapy or other biologic therapy) for lung cancer
* Patients must not have received prior chest radiation therapy for NSCLC
* Patients must not have had a previous surgical resection; however, patients may have undergone exploratory thoracotomy, mediastinoscopy, excisional biopsy or similar surgery for the purpose of determining the diagnosis, stage or potential resectability of newly diagnosed lung tumor; at least 28 days must have elapsed since thoracic surgery (excluding mediastinoscopy or other minor surgeries) and patients should have recovered from all associated toxicities at the time of registration; patients must not be planning to undergo a minor surgical procedure while on this study
* Patients must have Zubrod performance status 0-1
* Patients must have tumor tissue available for submission to assess gene expression of ERCC1 and XRCC1; patients must also be offered participation in banking for future use of specimens
* Absolute neutrophil count >= 1,500/mcl
* Platelets >= 100,000/mcl
* Hemoglobin >= 9.0 g/dl
* Total bilirubin within institutional upper limit of normal (IULN)
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) or serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 2.5 x IULN
* Patients must not be pregnant or nursing; women/men of reproductive potential must have agreed to use an effective contraceptive method; a woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months; in addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation; however, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures
* Patients must have a serum creatinine =< the IULN AND measured or calculated creatinine clearance >= 60 cc/min using the Cockroft-Gault formula
* Patients must have pulmonary function tests (PFTs) including forced expiratory volume in 1 second (FEV1) within 84 days prior to registration; for FEV1, the best value obtained pre- or post-bronchodilator must be >= 1.2 liters/second and/or >= 50% predicted
* Patients may not be planning to receive any other investigational agents
* Patients must not have more than 10% weight loss in the past 6 months
* Patients must not have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to ABT-888, carboplatin, paclitaxel or other agents used in study
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for five years
* Patient must not have any uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients must not currently have a > grade 1 symptomatic neuropathy-sensory (National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] version 4.0)
* Patients must not have a history of seizures
* Patients must not have any known immune deficiencies; patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy; therefore, known human immunodeficiency virus (HIV) positive patients receiving combination anti-retroviral therapy are excluded from the study
* Patients must be able to swallow whole capsules
* Prestudy history and physical must be obtained within 28 days prior to registration
* All patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* As a part of the Oncology Patient Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system
* REGISTRATION #2 - PRIOR TO CONSOLIDATION CHEMOTHERAPY:
* REGISTRATION #2 - PRIOR TO CONSOLIDATION CHEMOTHERAPY: Patients must have completed chemoradiotherapy per protocol and at least four weeks but no more than six weeks must have elapsed from the last day of induction therapy (the last day of radiation)
* REGISTRATION #2 - PRIOR TO CONSOLIDATION CHEMOTHERAPY: Patients must have undergone restaging tests according to the study calendar and determined to have no evidence of disease progression
* REGISTRATION #2 - PRIOR TO CONSOLIDATION CHEMOTHERAPY: Patients must have a serum creatinine =< (IULN) AND measured of calculated creatinine clearance >= 60 cc/min using the Cockroft-Gault formula
* REGISTRATION #2 - PRIOR TO CONSOLIDATION CHEMOTHERAPY: Absolute neutrophil count >= 1,500 mcl
* REGISTRATION #2 - PRIOR TO CONSOLIDATION CHEMOTHERAPY: Platelets >= 100,000/mcl
* REGISTRATION #2 - PRIOR TO CONSOLIDATION CHEMOTHERAPY: Hemoglobin >= 9.0 g/dl
* REGISTRATION #2 - PRIOR TO CONSOLIDATION CHEMOTHERAPY: Total bilirubin =< IULN
* REGISTRATION #2 - PRIOR TO CONSOLIDATION CHEMOTHERAPY: SGOT (AST) or SGPT (ALT) =< 2.5 x IULN
* REGISTRATION #2 - PRIOR TO CONSOLIDATION CHEMOTHERAPY: Patients must have Zubrod performance status 0-1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2011-06-20 (Actual); Primary Completion 2019-05-26 (Actual); Study Completion 2025-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Athanassios (Ethan) Argiris, Principal Investigator — SWOG Cancer Research Network
Locations (234):
- United States (234):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Tower Cancer Research Foundation, Beverly Hills, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - City of Hope Corona, Corona, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Mercy Cancer Center, Merced, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - OSF Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Reid Health, Richmond, Indiana
  - McFarland Clinic - Ames, Ames, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Saint Catherine Hospital, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - HaysMed, Hays, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - University of Kansas Cancer Center-West, Kansas City, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Bronson Battle Creek, Battle Creek, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Mercy Oncology and Hematology - Clayton-Clarkson, Ballwin, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - Kansas City Veterans Affairs Medical Center, Kansas City, Missouri
  - The University of Kansas Cancer Center-South, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - ECU Health Oncology Kinston, Kinston, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Cleveland Clinic Mercy Hospital, Canton, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC - Englewood, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Dayton Physicians LLC-Signal Point, Middletown, Ohio
  - Dayton Physicians LLC-Wilson, Sidney, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Dayton Physicians LLC - Troy, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Penn State Health Saint Joseph Medical Center, Reading, Pennsylvania
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - M D Anderson Cancer Center, Houston, Texas
  - Audie L Murphy VA Hospital, San Antonio, Texas
  - Cancer Therapy and Research Center at The UT Health Science Center at San Antonio, San Antonio, Texas
  - University Hospital, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Downtown, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - North, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Valley, Spokane Valley, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In phase I, 21 participants were enrolled (8 on 40mg cohort, 7 on 80mg cohort and 6 on 120mg cohort separately). All 21 participants met the eligibility criterial. 14 of 21 participants later went on to consolidation therapy.
  In phase II, 32 participants were enrolled. 1 was ineligible and thus excluded from analysis. 18 of 31 eligible participants were randomized to veliparib arm and 13 participants to the placebo arm. 23 of 31 eligible participants later on went on to consolidation therapy
Groups:
- Phase I 40 mg Veliparib Cohort: Participants undergo 3D-CRT and receive 40 mg veliparib, carboplatin, and paclitaxel during RT
- Phase I Consolidation 40mg Cohort; Phase I Consolidation 80mg Cohort; Phase I Consolidation 120mg Cohort: Participants receive 80 mg veliparib (PO twice daily, Days 1-7, Days 22-28), carboplatin, and paclitaxel for 2 cycles
- Phase I 80 mg Veliparib Cohort: Participants undergo 3D-CRT and receive 80 mg veliparib, carboplatin, and paclitaxel during RT
- Phase I 120 mg Veliparib Cohort: Participants undergo 3D-CRT and receive 120 mg veliparib, carboplatin, and paclitaxel during RT.
- Phase II Arm I (RT, Veliparib, Carboplatin, Paclitaxel): Participants undergo 3D-CRT and receive 120mg veliparib, carboplatin, and paclitaxel
  During consolidation, participants receive 80 mg veliparib (PO twice daily, Days 1-7, Days 22-28), carboplatin, and paclitaxel for 2 cycles.
- Phase II Arm II (3D-CRT, Placebo, Carboplatin, Paclitaxel): Participants undergo 3D-CRT and receive placebo PO BID, carboplatin and paclitaxel.
  During consolidation, participants receive 80 mg placebo (PO twice daily, Days 1-7, Days 22-28), carboplatin, and paclitaxel for 2 cycles.
Period: Phase I 40mg: Concurrent CRT
Arm/Group | Phase I 40 mg Veliparib Cohort | Phase I Consolidation 40mg Cohort | Phase I 80 mg Veliparib Cohort | Phase I Consolidation 80mg Cohort | Phase I 120 mg Veliparib Cohort | Phase I Consolidation 120mg Cohort | Phase II Arm I (RT, Veliparib, Carboplatin, Paclitaxel) | Phase II Arm II (3D-CRT, Placebo, Carboplatin, Paclitaxel)
Started | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Progression/relapse | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other- not protocol specified | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase I 40mg: Consolidation Therapy
Arm/Group | Phase I 40 mg Veliparib Cohort | Phase I Consolidation 40mg Cohort | Phase I 80 mg Veliparib Cohort | Phase I Consolidation 80mg Cohort | Phase I 120 mg Veliparib Cohort | Phase I Consolidation 120mg Cohort | Phase II Arm I (RT, Veliparib, Carboplatin, Paclitaxel) | Phase II Arm II (3D-CRT, Placebo, Carboplatin, Paclitaxel)
Started | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase I 80mg: Concurrent CRT
Arm/Group | Phase I 40 mg Veliparib Cohort | Phase I Consolidation 40mg Cohort | Phase I 80 mg Veliparib Cohort | Phase I Consolidation 80mg Cohort | Phase I 120 mg Veliparib Cohort | Phase I Consolidation 120mg Cohort | Phase II Arm I (RT, Veliparib, Carboplatin, Paclitaxel) | Phase II Arm II (3D-CRT, Placebo, Carboplatin, Paclitaxel)
Started | 0 | 0 | 7 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Period: Phase I 80mg: Consolidation Therapy
Arm/Group | Phase I 40 mg Veliparib Cohort | Phase I Consolidation 40mg Cohort | Phase I 80 mg Veliparib Cohort | Phase I Consolidation 80mg Cohort | Phase I 120 mg Veliparib Cohort | Phase I Consolidation 120mg Cohort | Phase II Arm I (RT, Veliparib, Carboplatin, Paclitaxel) | Phase II Arm II (3D-CRT, Placebo, Carboplatin, Paclitaxel)
Started | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase I 120mg: Concurrent CRT
Arm/Group | Phase I 40 mg Veliparib Cohort | Phase I Consolidation 40mg Cohort | Phase I 80 mg Veliparib Cohort | Phase I Consolidation 80mg Cohort | Phase I 120 mg Veliparib Cohort | Phase I Consolidation 120mg Cohort | Phase II Arm I (RT, Veliparib, Carboplatin, Paclitaxel) | Phase II Arm II (3D-CRT, Placebo, Carboplatin, Paclitaxel)
Started | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Refusal unrelated to AE | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: Phase I 120mg: Consolidation Therapy
Arm/Group | Phase I 40 mg Veliparib Cohort | Phase I Consolidation 40mg Cohort | Phase I 80 mg Veliparib Cohort | Phase I Consolidation 80mg Cohort | Phase I 120 mg Veliparib Cohort | Phase I Consolidation 120mg Cohort | Phase II Arm I (RT, Veliparib, Carboplatin, Paclitaxel) | Phase II Arm II (3D-CRT, Placebo, Carboplatin, Paclitaxel)
Started | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase II Concurrent CRT
Arm/Group | Phase I 40 mg Veliparib Cohort | Phase I Consolidation 40mg Cohort | Phase I 80 mg Veliparib Cohort | Phase I Consolidation 80mg Cohort | Phase I 120 mg Veliparib Cohort | Phase I Consolidation 120mg Cohort | Phase II Arm I (RT, Veliparib, Carboplatin, Paclitaxel) | Phase II Arm II (3D-CRT, Placebo, Carboplatin, Paclitaxel)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 18 | 13
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
Not completed — Refusal unrelated to AE | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Period: Phase II: Consolidation Therapy
Arm/Group | Phase I 40 mg Veliparib Cohort | Phase I Consolidation 40mg Cohort | Phase I 80 mg Veliparib Cohort | Phase I Consolidation 80mg Cohort | Phase I 120 mg Veliparib Cohort | Phase I Consolidation 120mg Cohort | Phase II Arm I (RT, Veliparib, Carboplatin, Paclitaxel) | Phase II Arm II (3D-CRT, Placebo, Carboplatin, Paclitaxel)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 13 | 10
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Not completed — Refusal unrelated to AE | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Progression/relapse | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: All eligible participants
Groups:
- Phase I 40mg Veliparib Cohort: Participants undergo 3D-CRT and receive 40 mg veliparib, carboplatin, and paclitaxel during RT 3-Dimensional Conformal Radiation Therapy: Undergo 3D-conformal RT Carboplatin: Given IV Laboratory Biomarker Analysis: Correlative studies Paclitaxel: Given IV Veliparib: Given PO
- Phase I 80mg Veliparib Cohort: Participants undergo 3D-CRT and receive 80 mg veliparib, carboplatin, and paclitaxel during RT 3-Dimensional Conformal Radiation Therapy: Undergo 3D-conformal RT Carboplatin: Given IV Laboratory Biomarker Analysis: Correlative studies Paclitaxel: Given IV Veliparib: Given PO
- Phase I 120mg Veliparib Cohort: Participants undergo 3D-CRT and receive 120 mg veliparib, carboplatin, and paclitaxel during RT 3-Dimensional Conformal Radiation Therapy: Undergo 3D-conformal RT Carboplatin: Given IV Laboratory Biomarker Analysis: Correlative studies Paclitaxel: Given IV Veliparib: Given PO
- Total: Total of all reporting groups
Arm/Group | Phase I 40mg Veliparib Cohort | Phase I 80mg Veliparib Cohort | Phase I 120mg Veliparib Cohort | Arm I (RT, Veliparib, Carboplatin, Paclitaxel) | Arm II (3D-CRT, Placebo, Carboplatin, Paclitaxel) | Total
Number analyzed (Participants) | 8 | 7 | 6 | 18 | 13 | 52
Age, Continuous [Median (Full Range); unit: years] | 69.2 [57.5 to 77.0] | 66.5 [61.4 to 80.9] | 69.7 [53.3 to 73.1] | 64.7 [47.0 to 78.9] | 65.0 [56.6 to 75.6] | 67.0 [47.0 to 80.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 1 | 11 | 6 | 24
  Male | 5 | 4 | 5 | 7 | 7 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 8 | 7 | 5 | 18 | 13 | 51
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 2 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 2 | 1 | 4
  White | 7 | 6 | 5 | 13 | 12 | 43
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 0 | 2
Zubrod Performance Status [Count of Participants; unit: Participants] — 0 - Fully active, able to carry on all pre-disease performance without restriction.
  1 - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work.
  Participants
    0 | 3 | 4 | 4 | 7 | 3 | 21
    1 | 5 | 3 | 2 | 11 | 10 | 31
Stage [Count of Participants; unit: Participants] — Tumors are staged per AJCC Cancer Staging Manual, 7th edition
  IIIA - T4 N0-1 M0 T3 N1 M0 T1-3 N2 M0
  IIIB - T4 N2 M0 T1-4 N3 M0
  Participants
    IIIA | 5 | 5 | 6 | 7 | 5 | 28
    IIIB | 3 | 2 | 0 | 11 | 8 | 24
Histology [Count of Participants; unit: Participants]
  Squamous cell | 3 | 3 | 2 | 10 | 5 | 23
  Adenocarcinoma | 5 | 4 | 3 | 8 | 8 | 28
  Other | 0 | 0 | 1 | 0 | 0 | 1
Baseline LDH [Count of Participants; unit: Participants] — LDH- lactate dehydrogenase
  Participants
    Normal | 4 | 5 | 6 | 16 | 9 | 40
    Elevated | 1 | 2 | 0 | 2 | 3 | 8
    Not reported | 3 | 0 | 0 | 0 | 1 | 4
Smoking Status [Count of Participants; unit: Participants]
  Current smoker | 1 | 0 | 3 | 8 | 6 | 18
  Former status | 6 | 6 | 1 | 9 | 7 | 29
  Never smoker | 1 | 1 | 2 | 1 | 0 | 5
Weight loss past 6 months [Count of Participants; unit: Participants]
  <5% | 3 | 6 | 6 | 14 | 8 | 37
  5%-10% | 5 | 1 | 0 | 4 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Veliparib When Given Concurrently With Standard Carboplatin/Paclitaxel and Radiotherapy, Determined According to Incidence of Dose Limiting Toxicity (DLT) (Phase I)
Description: DLTs will be graded using National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0. DLTs must be attributable (probably, possibly, definitely related) to the study regimen and only occur during RT or 2 weeks after completing RT.
  DLTs are defined as:
  1. Radiation esophagitis or dermatitis radiation Grade 3 that lasts > 7 consecutive days or Grade 4
  2. Grade 4 neutropenia for > 7 days or neutropenic fever ( ANC <500 and temperature >= 38.5 oC)
  3. Grade 4 thrombocytopenia
  4. Grade 4 nausea/vomiting despite appropriate antiemetic therapy
  5. Delays in radiotherapy or chemotherapy or ABT-888 due to toxicity of > 3 weeks
  6. All other non-hematologic toxicities >= Grade 3, except
     * anorexia
     * fatigue
     * infection without neutropenia
     * Grade 3 AST/ALT elevations <= 7 days, infusion reactions
     * Grade 3 or 4 lymphopenia
     * Grade 3 or 4 electrolyte abnormalities that are corrected to <=Grade 2 in < 48 hours
     * Grade 3 dehydration lasting < 7 days
Time Frame: 9 weeks
Population: Eligible participants evaluable for dose limiting toxicity assessment
Measure: Number; unit: dose limiting toxicity
Groups:
- Phase I 40mg Veliparib: During induction, participants undergo 3D-CRT and receive 40 mg veliparib (PO twice daily), carboplatin, and paclitaxel for 6 weeks.
  During consolidation, participants receive 40 mg veliparib (PO twice daily, Days 1-7, Days 22-28), carboplatin, and paclitaxel for 2 cycles.
- Phase I 80mg Veliparib: During induction, participants undergo 3D-CRT and receive 80mg veliparib (PO twice daily), carboplatin, and paclitaxel for 6 weeks.
  During consolidation, participants receive 80 mg veliparib (PO twice daily, Days 1-7, Days 22-28), carboplatin, and paclitaxel for 2 cycles.
- Phase I 120mg Veliparib: During induction, participants undergo 3D-CRT and receive 120mg veliparib (PO twice daily), carboplatin, and paclitaxel for 6 weeks.
  During consolidation, participants receive 120 mg veliparib (PO twice daily, Days 1-7, Days 22-28), carboplatin, and paclitaxel for 2 cycles.
Arm/Group | Phase I 40mg Veliparib | Phase I 80mg Veliparib | Phase I 120mg Veliparib
Number analyzed (Participants) | 6 | 6 | 5
dose limiting toxicity | 1 | 1 | 0

2. Primary Outcome: Progression-free Survival of Patients Treated With Chemoradiotherapy Plus Veliparib (Phase II)
Description: Time from date of registration to date of first documentation of progression or symptomatic deterioration or death due to any cause. Participants last known to be alive are censored at date of last contact.
  Assessed by Response Evaluation Criteria in Solid Tumors, RECIST 1.1
Time Frame: The time from randomization to progression or death due to any cause, assessed up to 5 years
Population: All eligible participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (RT, Veliparib, Carboplatin, Paclitaxel) | Arm II (3D-CRT, Placebo, Carboplatin, Paclitaxel)
Number analyzed (Participants) | 18 | 13
months | 9.3 [7.3 to 17.4] | 9.9 [5.7 to 23.6]

3. Secondary Outcome: Overall Survival (Phase II)
Description: From date of registration to date of death due to any cause. Participants last known to be alive are censored at date of last contact.
Time Frame: Up to 5 years
Population: All eligible participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (RT, Veliparib, Carboplatin, Paclitaxel) | Arm II (3D-CRT, Placebo, Carboplatin, Paclitaxel)
Number analyzed (Participants) | 18 | 13
months | 27.6 [17.4 to 27.6] | 15.2 [6.6 to 20.6]

4. Secondary Outcome: Objective Response Rate (Phase II)
Description: ORR is defined as the percentage of participants with evidence of a confirmed complete response (CR) or partial response (PR) as per Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1
Time Frame: Up to 5 years
Population: All eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (RT, Veliparib, Carboplatin, Paclitaxel) | Arm II (3D-CRT, Placebo, Carboplatin, Paclitaxel)
Number analyzed (Participants) | 18 | 13
percentage of participants | 56 [31 to 78] | 69 [38 to 91]

5. Secondary Outcome: Incidence of Serious (>= Grade 3) Adverse Events as Measured by National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0 (Phase II)
Description: Adverse Events (AEs) are reported by CTCAE Version 4.0. Only adverse events that are possibly, probably or definitely related to study drug are reported.
Time Frame: Duration of treatment and follow up until death or 5 years post registration
Population: Up to 4 weeks after completion of consolidation therapy
Measure: Number; unit: Participants
Groups:
- Arm I Concurrent Chemoradiation (Veliparib, 3D-CRT, Carboplati: Participants undergo 3D-CRT and receive veliparib, carboplatin, and paclitaxel as in Phase I induction and consolidation therapy.
  3-Dimensional Conformal Radiation Therapy: Undergo 3D-conformal RT Carboplatin: Given IV Laboratory Biomarker Analysis: Correlative studies Paclitaxel: Given IV Veliparib: Given PO
- Arm II Concurrent Chemoradiation (Placebo, 3D-CRT, Carboplatin: Participants undergo 3D-CRT as in arm I. Patients also receive placebo PO BID on days 1-43 and carboplatin and paclitaxel as in Phase I. Within 4-6 weeks after completion of chemotherapy and radiation therapy, participants receive placebo on days 1-7 and carboplatin and paclitaxel as in Phase I.
  3-Dimensional Conformal Radiation Therapy: Undergo 3D-conformal RT Carboplatin: Given IV Laboratory Biomarker Analysis: Correlative studies Paclitaxel: Given IV Placebo Administration: Given PO
- Arm I Consolidation (Veliparib, Carboplatin, Paclitaxel): Participants receive 80 mg veliparib (PO twice daily, Days 1-7, Days 22-28), carboplatin, and paclitaxel for 2 cycles.
- Arm II Consolidation (Placebo, Carboplatin, Paclitaxel): Participants receive 80mg placebo (PO twice daily, Days 1-7, Days 22-28), carboplatin, and paclitaxel for 2 cycles.
Arm/Group | Arm I Concurrent Chemoradiation (Veliparib, 3D-CRT, Carboplati | Arm II Concurrent Chemoradiation (Placebo, 3D-CRT, Carboplatin | Arm I Consolidation (Veliparib, Carboplatin, Paclitaxel) | Arm II Consolidation (Placebo, Carboplatin, Paclitaxel)
Number analyzed (Participants) | 17 | 13 | 12 | 10
Participants
  Anemia | 1 | 0 | 1 | 0
  Anorexia | 1 | 1 | 1 | 0
  Dehydration | 0 | 1 | 1 | 0
  Diarrhea | 0 | 0 | 1 | 0
  Dysphagia | 0 | 0 | 2 | 0
  Esophageal pain | 1 | 0 | 0 | 0
  Esophagitis | 1 | 1 | 0 | 0
  Fatigue | 1 | 1 | 1 | 0
  Hyperglycemia | 1 | 0 | 0 | 1
  Hypocalcemia | 0 | 1 | 0 | 0
  Hypoglycemia | 0 | 1 | 0 | 0
  Hypokalemia | 0 | 1 | 0 | 1
  Hypomagnesemia | 0 | 1 | 0 | 1
  Hyponatremia | 0 | 3 | 0 | 0
  Hypotension | 1 | 0 | 0 | 0
  Lung infection | 0 | 1 | 0 | 0
  Lymphocyte count decreased | 3 | 4 | 2 | 2
  Mucositis oral | 1 | 0 | 0 | 0
  Nausea | 0 | 0 | 1 | 0
  Neutrophil count decreased | 3 | 1 | 3 | 0
  Platelet count decreased | 1 | 0 | 1 | 0
  Pneumonitis | 0 | 1 | 0 | 1
  Upper gastrointestinal hemorrhage | 0 | 0 | 1 | 0
  Vomiting | 0 | 1 | 1 | 0
  Weight loss | 1 | 0 | 0 | 1
  White blood cell decreased | 2 | 2 | 2 | 0

ADVERSE EVENTS:
Time Frame: Duration of treatment and follow up until death or 5 years post registration
Description: Adverse Events (AEs) are reported by CTCAE Version 4.0.
  21 participants in phase I and 31 participants in phase II who were eligible and received protocol therapy were assessed for AEs. 1 participant in phase II arm 1 did not receive protocol therapy so was not assessed for AEs. All cause modality analysis will include all eligible participants as participants at risk.
Groups:
- Phase I 40 mg Veliparib Cohort: Participants undergo 3D-CRT and receive 40 mg veliparib, carboplatin, and paclitaxel during concurrent radiotherapy
- Phase I 80 mg Veliparib Cohort: Participants undergo 3D-CRT and receive 80 mg veliparib, carboplatin, and paclitaxel during concurrent radiotherapy
- Phase I 120 mg Veliparib Cohort; Phase II Arm I (Veliparib, 3D-CRT, Carboplatin, Paclitaxel): Participants undergo 3D-CRT and receive 120 mg veliparib, carboplatin, and paclitaxel during concurrent radiotherapy
- Phase II Arm II (Placebo, 3D-CRT, Carboplatin, Paclitaxel): Participants undergo 3D-CRT and receive placebo, carboplatin, and paclitaxel during concurrent radiotherapy
- Phase II Arm I Consolidation: Participants receive 80 mg veliparib (PO twice daily, Days 1-7, Days 22-28), carboplatin, and paclitaxel for 2 cycles.
- Phase II Arm II Consolidation: Participants receive 80 mg placebo (PO twice daily, Days 1-7, Days 22-28), carboplatin, and paclitaxel for 2 cycles.
Arm/Group | Phase I 40 mg Veliparib Cohort | Phase I 80 mg Veliparib Cohort | Phase I 120 mg Veliparib Cohort | Phase II Arm I (Veliparib, 3D-CRT, Carboplatin, Paclitaxel) | Phase II Arm II (Placebo, 3D-CRT, Carboplatin, Paclitaxel) | Phase I Consolidation 40mg Cohort | Phase I Consolidation 80mg Cohort | Phase I Consolidation 120mg Cohort | Phase II Arm I Consolidation | Phase II Arm II Consolidation
All-Cause Mortality (participants affected / at risk) | 7/8 | 5/7 | 2/6 | 8/18 | 8/13 | 3/4 | 3/5 | 2/5 | 7/13 | 6/10
Serious Adverse Events (participants affected / at risk) | 3/8 | 3/7 | 2/6 | 2/17 | 3/13 | 1/4 | 0/5 | 1/5 | 3/12 | 1/10
Other Adverse Events (participants affected / at risk) | 8/8 | 7/7 | 6/6 | 17/17 | 13/13 | 4/4 | 4/5 | 5/5 | 12/12 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I 40 mg Veliparib Cohort (N=8) | Phase I 80 mg Veliparib Cohort (N=7) | Phase I 120 mg Veliparib Cohort (N=6) | Phase II Arm I (Veliparib, 3D-CRT, Carboplatin, Paclitaxel) (N=17) | Phase II Arm II (Placebo, 3D-CRT, Carboplatin, Paclitaxel) (N=13) | Phase I Consolidation 40mg Cohort (N=4) | Phase I Consolidation 80mg Cohort (N=5) | Phase I Consolidation 120mg Cohort (N=5) | Phase II Arm I Consolidation (N=12) | Phase II Arm II Consolidation (N=10)
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Esophageal perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Esophagitis (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Death NOS (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight loss (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intracranial hemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vasovagal reaction (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Thromboembolic event (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I 40 mg Veliparib Cohort (N=8) | Phase I 80 mg Veliparib Cohort (N=7) | Phase I 120 mg Veliparib Cohort (N=6) | Phase II Arm I (Veliparib, 3D-CRT, Carboplatin, Paclitaxel) (N=17) | Phase II Arm II (Placebo, 3D-CRT, Carboplatin, Paclitaxel) (N=13) | Phase I Consolidation 40mg Cohort (N=4) | Phase I Consolidation 80mg Cohort (N=5) | Phase I Consolidation 120mg Cohort (N=5) | Phase II Arm I Consolidation (N=12) | Phase II Arm II Consolidation (N=10)
Anemia (Blood and lymphatic system disorders) | 6 | 3 | 3 | 8 | 10 | 3 | 1 | 2 | 5 | 9
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac disorders-Other (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chest pain - cardiac (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mobitz (type) II atrioventricular block (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Paroxysmal atrial tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 2 | 1 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 2
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Blurred vision (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye disorders-Other (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 3
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 2 | 3 | 6 | 4 | 0 | 1 | 0 | 2 | 2
Diarrhea (Gastrointestinal disorders) | 2 | 2 | 2 | 6 | 1 | 0 | 0 | 1 | 2 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 3 | 1 | 2 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 2 | 3 | 6 | 5 | 0 | 1 | 1 | 4 | 3
Esophageal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Esophagitis (Gastrointestinal disorders) | 5 | 4 | 4 | 8 | 8 | 3 | 1 | 2 | 1 | 3
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Hemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 4 | 3 | 3 | 8 | 8 | 2 | 1 | 1 | 2 | 5
Stomach pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 2 | 5 | 4 | 0 | 0 | 0 | 2 | 1
Chills (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Edema limbs (General disorders) | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 2
Fatigue (General disorders) | 4 | 4 | 5 | 14 | 8 | 2 | 1 | 3 | 8 | 8
Fever (General disorders) | 0 | 1 | 0 | 3 | 2 | 0 | 0 | 0 | 2 | 0
General disorders and admin site conditions - Other (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 3 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 1 | 0
Allergic reaction (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchial infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Esophageal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Mucosal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Papulopustular rash (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Upper respiratory infection (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis radiation (Injury, poisoning and procedural complications) | 3 | 4 | 2 | 3 | 3 | 0 | 0 | 0 | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 1
Alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 3
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
CD4 lymphocytes decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac troponin I increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholesterol high (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Creatinine increased (Investigations) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
INR increased (Investigations) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Investigations-Other (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 6 | 5 | 4 | 7 | 9 | 2 | 2 | 2 | 2 | 6
Neutrophil count decreased (Investigations) | 3 | 4 | 3 | 6 | 2 | 1 | 4 | 0 | 4 | 1
Platelet count decreased (Investigations) | 3 | 1 | 4 | 5 | 4 | 1 | 2 | 1 | 5 | 2
Weight gain (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight loss (Investigations) | 3 | 1 | 0 | 5 | 3 | 1 | 0 | 0 | 3 | 3
White blood cell decreased (Investigations) | 6 | 5 | 3 | 6 | 8 | 1 | 3 | 1 | 3 | 2
Anorexia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 5 | 4 | 1 | 1 | 0 | 3 | 2
Dehydration (Metabolism and nutrition disorders) | 2 | 1 | 1 | 2 | 3 | 0 | 0 | 0 | 1 | 0
Glucose intolerance (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 2 | 2 | 3 | 5 | 0 | 0 | 0 | 1 | 3
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypernatremia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 1 | 0 | 3 | 7 | 1 | 0 | 1 | 2 | 4
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 3 | 1 | 0 | 1 | 3 | 1 | 0 | 1 | 0 | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 1 | 4 | 1 | 0 | 0 | 1 | 4
Hyponatremia (Metabolism and nutrition disorders) | 4 | 1 | 2 | 3 | 8 | 1 | 0 | 1 | 1 | 1
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 3 | 0 | 2 | 0 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 2
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 3
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 1 | 0 | 4 | 4 | 2 | 1 | 0 | 2 | 2
Dysgeusia (Nervous system disorders) | 1 | 4 | 0 | 1 | 2 | 0 | 2 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 1 | 6 | 0 | 0 | 0 | 0 | 3
Hypersomnia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Paresthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 0 | 2 | 3 | 1 | 2 | 1 | 3 | 2
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Confusion (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 1 | 1 | 2 | 0 | 0 | 0 | 2 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary frequency (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Urinary tract pain (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 3 | 6 | 2 | 0 | 0 | 0 | 2 | 5
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 1 | 3 | 4 | 0 | 0 | 0 | 2 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 2 | 3 | 3 | 0 | 0 | 0 | 2 | 1
Resp, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 0
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 4 | 1 | 2 | 1 | 2 | 5 | 6
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 2 | 0 | 2 | 2 | 0 | 1 | 0 | 0 | 1
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 2 | 1 | 1 | 3 | 0 | 1 | 0 | 0 | 2
Hypotension (Vascular disorders) | 3 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0
Thromboembolic event (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-12): https://cdn.clinicaltrials.gov/large-docs/85/NCT01386385/Prot_SAP_000.pdf